CLINICAL TRIAL: NCT02020070
Title: A Phase 2 Study Combining Ipilimumab, Degarelix, and Radical Prostatectomy in Men With Newly Diagnosed Metastatic Castration Sensitive Prostate Cancer or Ipilimumab and Degarelix in Men With Biochemically Recurrent Castration Sensitive Prostate Cancer After Radical Prostatectomy
Brief Title: Combining Ipilimumab, Degarelix, and Radical Prostatectomy in Men With Newly Diagnosed Metastatic Castration Sensitive Prostate Cancer or Ipilimumab and Degarelix in Men With Biochemically Recurrent Castration Sensitive Prostate Cancer After Radical Prostatectomy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-134
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Castration Sensitive Prostate Cancer
Keywords: Ipilimumab; Degarelix; Radical Prostatectomy; 13-134
MeSH Terms: interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Ipilimumab

ARMS (2):
- Ipilimumab & Degarelix With Radical Prostatectomy (Experimental): Week 1: Degarelix SQ injection (except patients who have already received hormonal therapy per standard of care and are not yet due for their next dose) and Ipilimumab at 3 mg/kg intravenously (IV). Surgery Radical prostatectomy (RP)will be performed during week 3 ± 1 week or after recovery to grade ≤ 1 adverse events experienced during the induction period related to treatment. Continued Androgen Depletion and Ipilimumab Weeks 5, 9, 13, 17, 21, 25, and 29: Degarelix 80 mg SQ (except patients who have already received hormonal therapy per standard of care and are not yet due for their next dose)
  Week 11, 14, 17 or after sufficient wound healing and recovery post RP:
  Ipilimumab 3 mg/kg IV Follow-up Twelve week intervals until Week 87.
  Interventions: Drug: Degarelix; Drug: Ipilimumab; Procedure: Radical Prostatectomy
- Ipilimumab & Degarelix With Prior With Radical Prostatectomy (Experimental): Week 1: Degarelix 240 mg SQ injection and Ipilimumab at 3 mg/kg intravenously (IV) Continued Androgen Depletion and Ipilimumab Weeks 5, 9, 13, 17, 21, 25, and 29: Degarelix 80 mg SQ Week 4,7,10: Ipilimumab 3mg/kg IV Follow-up Twelve week intervals until Week 81, with MD visits at weeks 52 and 84 (12 and 20 months).
  Interventions: Drug: Degarelix; Drug: Ipilimumab

INTERVENTIONS:
Drug: Degarelix
Drug: Ipilimumab
Procedure: Radical Prostatectomy
  Arms: Ipilimumab & Degarelix With Radical Prostatectomy

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, taking ipilimumab with degarelix before surgery to remove the prostate, followed by more degarelix and ipilimumab after the surgery, will have on prostate cancer.

The goal of this trial is to assess the safety and efficacy of a multimodality approach combining hormones and immunotherapy in prostate cancer populations that are considered incurable and standardly treated with hormones alone, and represent clinical states prior to development of castration-resistant disease. There are 2 cohorts. The first will use ipilimumab and degarelix prior to and following radical prostatectomy in men with newly diagnosed, oligometastatic, castration-sensitive disease. The second cohort will include men who have already received definitive local therapy with radical prostatectomy but have since experienced biochemical and/or metastatic recurrence.

ELIGIBILITY:
Inclusion Criteria:

Target Population: Cohort A Patients with castration-sensitive oligometastatic prostate cancer who have not received primary local therapy (radiation or surgery), and no more than 5 months of prior androgen deprivation therapy.

* The subject must be age 18 or older, and be willing and able to provide informed consent.
* The subject must have histologically confirmed adenocarcinoma of the prostate with tissue confirmation at selected study site.
* The subject must have newly diagnosed prostate cancer with a metastatic site(s).
* The subject must have a history or presence of ≤ 10 bony metastatic lesions
* Note: bone mets that are not clearly identified on bone imaging, but are biopsy proven are allowed
* History or presence of distant metastatic lymph node(s) (e.g., retroperitoneal or non-regional pelvic lymph nodes) are allowed
* History or presence of regional pelvic lymph nodes (as per AJCC Cancer Staging [7th edition]) will be considered a metastatic site if greater than 1.5cm in shortest dimension.
* The subject must have Karnofsky performance status of 80-100.
* Normal organ function with acceptable initial laboratory values:

  * WBC ≥ 2000/μL
  * ANC ≥ 1000/ μL
  * Platelets ≥ 75 x 103/μL
  * Creatinine ≤ 2.0 x ULN
  * AST/ALT ≤ 2.5 x ULN
  * Bilirubin ≤ 1.5 x ULN (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* No active or chronic infection with HIV, Hepatitis B or Hepatitis C (negative screening tests required).
* The subject must be deemed medically fit for radical prostatectomy by the attending urologic surgeon at the selected study site.
* Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study [and for up to 26 weeks after the last dose of ipilimumab] in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* Patients that meet any of the criteria listed below will not be eligible for Cohort A entry:
* Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer or superficial bladder cancer
* Major surgery within 4 weeks of enrollment (Week 1 Visit).
* Current or prior radiation therapy to the prostate Prior radiation to a metastatic site (e.g., palliative radiation) is allowed..
* More than 5 months of prior hormonal therapy (e.g., gonadotropin hormone releasing analogs, megestrol acetate, or casodex) . There is no washout period required for GnRH analogs. A two week washout is required for megestrol or anti-androgen.
* Prior use of an 5 alpha reductase inhibitor is allowed (no limit on duration of use), however a two week washout is required.
* Prior ketoconazole, abiraterone acetate, or enzalutamide for the treatment of prostate cancer.
* Current or prior investigational therapies for prostate cancer, or chemotherapy administered with the intent to treat prostate cancer.
* Concomitant therapy with any other experimental drug.
* Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]); motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis).
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
* Patients with underlying heart conditions who are deemed ineligible for surgery.
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab).
* Note: Inactivated vaccines are allowed at any time on study.
* A history of prior treatment with ipilimumab or prior CD137 agonist or CTLA-4 inhibitor or agonist.
* Concomitant or prior therapy with any of the following: IL-2, interferon, or other nonstudy immunotherapy regimens; immunosuppressive agents; ; or chronic use of systemic corticosteroids within 6 weeks of study entry.
* Persons of reproductive potential unwilling to use an adequate method of contraception throughout treatment and for at least 26 weeks after ipilimumab is stopped.
* Patients who have had a history of acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation.

Inclusion Criteria:

Target Population: Cohort B

* The subject must be age 18 or older, and be willing and able to provide informed consent.
* Histologically confirmed prostate cancer with progressive disease, defined as:
* Rising PSA (50% or more increase to a level of 1 ng/mL or more, based on at least 3 PSA determinations obtained at least 1 week apart). The 50% rise in PSA is across the 3 determinations, and these determinations do not need to be sequential.
* PSA doubling time of ≤ 12 months as calculated according to the Memorial Sloan-Kettering Cancer Center nomogram (http://www.mskcc.org/mskcc/html/10088.cfm)

  * The subject must have Karnofsky performance status of 80-100.
  * Normal organ function with acceptable initial laboratory values:
  * WBC ≥ 2000/μL
  * ANC ≥ 1000/ μL
  * Platelets ≥ 75 x 103/μL
  * Creatinine ≤ 2.0 x ULN
  * AST/ALT ≤ 2.5 x ULN
  * Bilirubin ≤ 1.5 x ULN (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* No active or chronic infection with HIV, Hepatitis B or Hepatitis C (negative screening tests required).
* Prior radiotherapy to the prostate (adjuvant or salvage radiotherapy) is allowed
* Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study [and for up to 26 weeks after the last dose of ipilimumab] in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

Target Population: Cohort B

Patients that meet any of the criteria listed below will not be eligible for Cohort B entry:

* Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer or superficial bladder cancer
* Major surgery within 4 weeks of enrollment (Week 1 Visit).
* Visceral metastatic disease
* More than 3 cycles of intermittent hormones (for the treatment of biochemical recurrence or castration sensitive metastatic disease), with a cycle defined as a period of consistent androgen deprivation therapy (generally 3-12 months) followed by intentional cessation of ADT without reinitiation of ADT until the PSA rises.
* Prior use of an 5 alpha reductase inhibitor is allowed (no limit on duration of use), however a two week washout is required.
* Current or prior investigational therapies for prostate cancer, or chemotherapy administered with the intent to treat prostate cancer.
* Concomitant therapy with any other experimental drug.
* Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]); motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis).
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab).
* Note: Inactivated vaccines are allowed at any time on study.
* A history of prior treatment with ipilimumab or prior CD137 agonist or CTLA-4 inhibitor or agonist.
* Concomitant or prior therapy with any of the following: IL-2, interferon, or other non-study immunotherapy regimens; immunosuppressive agents; ; or chronic use of systemic corticosteroids within 6 weeks of study entry.
* Persons of reproductive potential unwilling to use an adequate method of contraception throughout treatment and for at least 26 weeks after ipilimumab is stopped.
* Patients who have had a history of acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
undetectable PSA | at 12 and 20 months
  An undetectable PSA at 12 and 20 months (weeks 52 and 84, respectively) from the start of treatment among patients with non-castrate (> 150 ng/ml) levels of testosterone. An undetectable PSA is defined as PSA ≤0.05 ng/mL.

SECONDARY OUTCOMES:
progression-free survival (PFS) | 2 years
  Progression-free survival (PFS) is a composite endpoint defined as disease progression in bone or soft-tissue, symptoms, or death measured from study entry. Progression in soft tissue will be measured by modified RECIST per PCWG2..
overall survival (OS) | 2 years
  Overall survival is defined as death from any cause measured from study entry.
Toxicity | 2 years
  Toxicity will be evaluated for all treated patients using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 (http://ctep.cancer.gov).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Autio, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/